CLINICAL TRIAL: NCT01239134
Title: Part A: A First-in-Human Single Ascending Dose Study of TRX518 in Subjects With Unresectable Stage III or Stage IV Malignant Melanoma or Other Solid Tumor Malignancies Part B: A Dose-Escalation Study of Multi-dose TRX518 Monotherapy Part C: An Expansion Cohort of Multi-dose TRX518 Monotherapy at the Maximum Tolerated Dose
Brief Title: Trial of TRX518 (Anti-GITR mAb) in Stage III or IV Malignant Melanoma or Other Solid Tumors
Acronym: TRX518-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leap Therapeutics, Inc. (Industry)
Collaborators: Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRX518-001
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Unresectable Stage III or Stage IV Malignant Melanoma or Other Solid Tumor Malignancies
Keywords: Malignant melanoma; Metastatic; Unresectable; Stage III or Stage IV; Solid tumor
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- TRX518 (Experimental)
  Interventions: Biological: TRX518

INTERVENTIONS:
Biological: TRX518 — Humanized, Fc disabled, anti-human GITR (glucocorticoid-induced tumor necrosis factor receptor) monoclonal antibody

SUMMARY:
TRX518-001 is an open label, non-randomized single group assignment, Phase 1 single dose escalation study in adults with biopsy proven unresectable Stage III or Stage IV melanoma or other solid tumor malignancies.

Part A: The study objectives are to determine the safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) profiles of TRX518 and to define the maximum tolerated dose at which there are tolerable side effects and/or maximum PK/PD parameter changes.

Subjects will be assigned to a cohort in the order screening is completed. Dose will depend upon the cohort in which a subject is enrolled and cohorts will be dosed consecutively by ascending dose. Part A has been completed.

Part B: A Dose-Escalation Study of Multi-dose TRX518 Monotherapy with objectives including characterization of the safety, tolerability, and pharmacokinetics, as well as, evaluate for evidence of anti-tumor activity and assess TRX518 immunogenicity.

Part C: An Expansion Cohort of Multi-dose TRX518 Monotherapy at the Maximum Tolerated Dose

DETAILED DESCRIPTION:
The following visits are required:

Part A:

* Screening visit: 1 to 2 appointments will be conducted to determine eligibility. All or most requirements can be determined from the patient's medical records.
* Baseline visit: within 7 days of the planned study dosing day a baseline physical exam, blood tests and electrocardiogram will be obtained.
* Dosing visit: 1 outpatient visit where TRX518 will be given IV over 1 hour followed by 4 hours of observation and some repeat blood tests.
* Follow up visits: 5 outpatient visits following dosing at 1, 8 and 15 days and 3, 6, 12, and 18 weeks post dosing
* Long term follow-up: 4 brief assessments by medical record review and/or telephone contact at 6, 12, 18, and 24 months post dosing.
* The core study duration is 18 weeks. The follow-up study duration is 24 months.

Parts B & C:

* Screening/Baseline visit: 1 appointment will be conducted to perform testing and evaluations for eligibility within 28 days of the first dosing day.
* Dosing Visits: Each subject will receive IV doses of TRX518 once every other week (e.g., D1 and D15) in 28-day cycles
* Follow up visits: When a patient stops treatment, they will enter the Follow-up Period and have an End of Treatment study visit approximately 30 days after the last dose of study drug. Subsequently, patients will have long-term follow-up approximately every 12 weeks until death or lost to follow up.

ELIGIBILITY:
Inclusion Criteria (Parts B & C):

* 18 years or older
* Histologically confirmed unresectable Stage III or Stage IV malignant melanoma, or other solid tumor malignancies
* Failed to respond to or relapsed following standard treatment, declined or was not eligible for standard treatment.
* Expected survival of at least 12 weeks.
* Eastern Cooperative Oncology Group performance status score of 0 or 1 is required.
* Evidence of adequate organ function by standard laboratory tests.

Exclusion Criteria (Parts B & C):

* Evidence of progression of central nervous system (CNS) metastases or symptomatic CNS metastases within 35 days prior to dosing.
* Ocular melanoma which has not metastasized or presence of a non-solid tumor.
* A history of any major surgery within 4 weeks prior to dosing.
* Any history of antitumor therapy completed within 28 days prior to dosing.
* Subjects with active autoimmune disease or history of known or suspected autoimmune disease, with the exception of subjects with isolated vitiligo, resolved childhood asthma/atopy, psoriasis not requiring systemic treatment and controlled thyroid disorders.
* Clinically significant heart disease, defined as NYHA Class III or IV.
* Any significant systemic infection requiring IV antibiotics.
* Known to be human immunodeficiency virus (HIV) positive, have hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCAb) unless HCV RNA undetected/negative.
* Treatment with any other anti-human GITR monoclonal antibody (mAb) or immunomodulatory therapy 42 days prior to dosing (30 days for Interleukin-2 & Interferon-α, 7 days for Topical Imiquimod).
* Adverse events from prior anti-cancer therapy that have not resolved to grade ≤1 except for alopecia, vitiligo, or endocrinopathy managed with replacement therapy.
* Use of any investigational drugs within 30 days prior to dosing.
* Any condition that requires or is likely to require treatment with pharmacologic doses of systemic corticosteroids. Subjects are permitted to receive physiologic replacement of corticosteroid therapy (≤ 10 mg prednisone daily).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Part A: Adverse Events | through 30 days post last dose
  Any adverse change in health or side effect from the initiation of the study drug dose through completion or premature withdrawal
Part A: TRX518 peak concentration (Cmax) | various timepoints through 1 week post dose
  Observations of the distribution, duration of effects and chemical changes of TRX518 in the body and the effects and routes of the body's elimination of TRX518
Part A: Time to peak concentration (Tmax) | various timepoints through 1 week post dose
  Observations of the distribution, duration of effects and chemical changes of TRX518 in the body and the effects and routes of the body's elimination of TRX518
Part A: Area under the curve (AUC) | various timepoints through 1 week post dose
  Observations of the distribution, duration of effects and chemical changes of TRX518 in the body and the effects and routes of the body's elimination of TRX518
Part A: Define a maximum single dose at which there are tolerable side effects and/or maximum PK/PcD parameter changes | End of Cycle 1 (Day 28)
Parts B and C: Adverse Events | through 30 days post dose
  Any adverse change in health or side effect from the initiation of the study drug dose through completion or premature withdrawal

SECONDARY OUTCOMES:
Part A: Evaluate the effect of TRX518 on lymphoid cell subset number and function | At baseline and at various timepoints up to 6 weeks post dose
Part A: Assess TRX518 immunogenicity | At baseline and at various timepoints up to 18 weeks post dose
Part A: Evaluate the effect of TRX518 on long-term safety measuring vital signs, tumor status, adverse events | At Months 6, 12, 18 and 24
Parts B & C: TRX518 peak concentration (Cmax) | At each study visit from baseline up to end of treatment visit
  Observations of the distribution, duration of effects and chemical changes of TRX518 in the body and the effects and routes of the body's elimination of TRX518
Parts B & C: Time to peak concentration (Tmax) | At each study visit from baseline up to end of treatment visit
  Observations of the distribution, duration of effects and chemical changes of TRX518 in the body and the effects and routes of the body's elimination of TRX518
Parts B & C: Area under the curve (AUC) | At each study visit from baseline up to end of treatment visit
  Observations of the distribution, duration of effects and chemical changes of TRX518 in the body and the effects and routes of the body's elimination of TRX518
Parts B & C: Evaluate multi-dose TRX18 monotherapy for any evidence of antitumor activity (objective response rate, [ORR] progression free survival [PFS], duration of response and overall survival [OS]; RECIST v1.1 will be utilized | Every 8 weeks while on study treatment and every 12 weeks for survival until death or lost to follow up.
  objective response rate [ORR], progression free survival [PFS], duration of response [DoR] and overall survival [OS]); RECIST v1.1 criteria will be utilized
Parts B & C: Evaluate the effect of multi-dose TRX518 monotherapy on lymphoid cell subset number and function | At baseline and at various timepoints up to end of treatment visit
Parts B & C: Assess TRX518 immunogenicity | At baseline and at various timepoints up to end of treatment visit

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Sirard, Study Director — Leap Therapeutics
Locations (1):
- Immunotherapeutics Core / Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Melanoma Trials at MSKCC — http://www.mskcc.org/mskcc/html/14327.cfm